CLINICAL TRIAL: NCT01640730
Title: An Open Label Safety and Exploratory Efficacy Study of Kanglaite Injection in Patients Having Progressive Stage IV NSCLC Who Are Not Candidates for Other Anti-cancer Treatment
Brief Title: Safety and Exploratory Efficacy of Kanglaite Injection in Non Small Cell Lung Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: poor enrollment
Sponsor: KangLaiTe USA (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KLT-NSCLC-004
Record Dates: First submitted 2012-06-15; First posted 2012-07-16 (Estimated); Last update posted 2014-01-16 (Estimated); Status verified 2014-01

CONDITIONS: Stage IV NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — kang-lai-te

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Kanglaite injection (Experimental)
  Interventions: Drug: Kanglaite Injection

INTERVENTIONS:
Drug: Kanglaite Injection — 30gm IV infusion 5 days a week for 3 weeks every 28 days
  Other Names: KLTi

SUMMARY:
This study is for patients with advanced non small cell lung cancer that has progressed despite standard of care. The purpose of the study is to see if Kanglaite injection has any effect on survival.

ELIGIBILITY:
Inclusion Criteria:

* confirmed (within last 3 months)progressive Stage IV NSCLC
* estimated life span of 3 months
* phase angle of at least 5 as measured by bioimpedance

Exclusion Criteria:

* currently taking a lipid lowering medications
* has an imminently life threatening condition
* has pre-existing liver disease
* known allergy to soybeans
* uncontrolled diabetes or uncontrolled disturbance of lipid metabolism
* pregnant or lactating
* has a pacemaker or other implantable electronic medical device

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2012-05; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Overall Survival | from date of enrollment until date of death from any cause assessed up to 12 months

SECONDARY OUTCOMES:
Bioimpedance Phase Angle | measured each month up to one year
Palliation Response Measure | each month up to one year
  quality of life survey and performance status

CONTACTS AND LOCATIONS:
Locations (1):
- The West Clinic, Memphis, Tennessee, United States